CLINICAL TRIAL: NCT05503264
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Basket Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab in Patients With Anti-N-methyl-D-aspartic Acid Receptor (NMDAR) or Anti-leucine-rich Glioma-inactivated 1 (LGI1) Encephalitis
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Satralizumab in Participants With Anti-N-methyl-D-aspartic Acid Receptor (NMDAR) or Anti-leucine-rich Glioma-inactivated 1 (LGI1) Encephalitis
Acronym: Cielo
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WN43174; 2021-002395-39 (EudraCT Number); 2023-504226-18-00 (EU CTIS Number)
Record Dates: First submitted 2022-08-15; First posted 2022-08-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: NMDAR Autoimmune Encephalitis; LGI1 Autoimmune Encephalitis
MeSH Terms: interventions — satralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NMDAR Autoimmune Encephalitis (AIE) Cohort (Experimental): Adults and adolescents with definite or probable NMDAR encephalitis
  Interventions: Drug: Satralizumab
- LGI1 AIE Cohort (Experimental): Adults with LGI1 encephalitis
  Interventions: Drug: Satralizumab
- NMDAR AIE Placebo Cohort (Placebo Comparator): Adults and adolescents with definite or probable NMDAR encephalitis
  Interventions: Other: Placebo
- LGI1 AIE Placebo Cohort (Placebo Comparator): Adults with LGI1 encephalitis
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Satralizumab — In Part 1, study drug will be administered after all other study-related procedures have been performed at a site visit at Weeks 0, 2, 4, and every 4 weeks (Q4W) thereafter. Participants will receive satralizumab according to body weight. Study drug will be administered by subcutaneous (SC) injection in the abdominal or femoral region after all other study-related procedures have been performed at a site visit. In Part 2, participants will be asked to choose from one of the following options: Option 1: continue on randomized, double-blind study drug; Option 2: start open-label satralizumab based on body weight; Option 3: stop study treatment and continue follow-up assessments.
  Arms: LGI1 AIE Cohort; NMDAR Autoimmune Encephalitis (AIE) Cohort
Other: Placebo — Satralizumab placebo prefilled syringe (PFS) is identical in composition to satralizumab PFS, but does not contain the satralizumab active ingredient and will be identical in appearance and packaging to satralizumab. A PFS (assembled with an needle safety device [NSD] and extended finger flange) filled with 0.5 milliliters (mL) of solution, corresponding to 60 milligrams (mg) satralizumab, may be used in Part 2 once it becomes available at the study site.
  Arms: LGI1 AIE Placebo Cohort; NMDAR AIE Placebo Cohort

SUMMARY:
The purpose of this study is to assess the efficacy, safety, PK, and PD of satralizumab in participants with NMDAR and LGI1 encephalitis.

ELIGIBILITY:
Inclusion Criteria:

* Reasonable exclusion of tumor or malignancy before baseline visit (randomization)
* Onset of AIE symptoms ≤ 9 months before randomization
* Meet the definition of "New Onset" or "Incomplete Responder" AIE
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate contraception during the treatment period and for at least 3 months after the final dose of satralizumab or placebo
* For participants enrolled in the extended China enrollment phase at China's sites: participants who are current residents of mainland China, Hong Kong, or Taiwan, and of Chinese ancestry

NMDAR AIE Cohort:

* Age ≥ 12 years
* Diagnosis of probable or definite NMDAR encephalitis

LGI1 AIE Cohort

* Age ≥ 18 years
* Diagnosis of LGI1 encephalitis

Exclusion Criteria:

* Any untreated teratoma or thymoma at baseline visit (randomization)
* History of carcinoma or malignancy, unless deemed cured by adequate treatment with no evidence of recurrence for ≥ 5 years before screening
* For participants with NMDAR AIE, history of negative anti-NMDAR antibody in cerebrospinal fluid (CSF) using a cell-based assay within 9 months of symptom onset
* Historically known positivity to an intracellular antigen with high cancer association or glutamate decarboxylase 65 (GAD-65)
* Historically known positivity to any cell surface neuronal antibodies other than NMDAR and LGI1, in the absence of NMDAR and LGI1 antibody positivity
* Confirmed paraneoplastic encephalitis
* Confirmed central or peripheral nervous system demyelinating disease
* Alternative causes of associated symptoms
* History of herpes simplex virus encephalitis in the previous 24 weeks
* Any previous/concurrent treatment with interleukin-6 (IL-6) inhibitory therapy (e.g., tocilizumab), alemtuzumab, total body irradiation, or bone marrow transplantation
* Any previous treatment with anti-cluster of differentiation 19 antibody (CD19 antibody), complement inhibitors, neonatal Fc receptor antagonists, anti-B-lymphocyte stimulator monoclonal antibody
* Any previous treatment with T-cell depleting therapies, cladribine, or mitoxantrone
* Treatment with oral cyclophosphamide within 1 year prior to baseline
* Treatment with any investigational drug (including bortezomib) within 24 weeks prior to screening
* Concurrent use of more than one immunosuppressive therapy (IST) as background therapy
* Contraindication to all of the following rescue treatments: rituximab, intravenous immunoglobulin (IVIG), high-dose corticosteroids, or intravenous (IV) cyclophosphamide
* Any surgical procedure, except laparoscopic surgery or minor surgeries within 4 weeks prior to baseline, excluding surgery for thymoma or teratoma removal
* Planned surgical procedure during the study
* Evidence of progressive multifocal leukoencephalopathy
* Evidence of serious uncontrolled concomitant diseases
* Congenital or acquired immunodeficiency, including human immunodeficiency virus (HIV) infection
* Active or presence of recurrent bacterial, viral, fungal, mycobacterial infection, or other infection
* Infection requiring hospitalization or treatment with IV anti-infective agents within 4 weeks prior to baseline visit
* Positive hepatitis B (HBV) and hepatitis C (HCV) test at screening
* Evidence of latent or active tuberculosis (TB)
* History of drug or alcohol abuse within 1 year prior to baseline
* History of diverticulitis or concurrent severe gastrointestinal (GI) disorders that, in the investigator's opinion, may lead to increased risk of complications such as GI perforation
* Receipt of live or live-attenuated vaccine within 6 weeks prior to baseline visit
* History of blood donation (1 unit or more), plasma donation or platelet donation within 90 days prior to screening
* History of severe allergic reaction to a biologic agent
* History of suicide attempt within 3 years prior to screening except if this is clearly associated with and occurs during the acute phase of LGI-1 or NMDAR encephalitis
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes safe participation in and completion of the study
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of study drug

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2029-12-14 (Estimated)

PRIMARY OUTCOMES:
Part 1: Proportion of Participants in NMDAR AIE Cohort With Modified Rankin Scale (mRS) Score Improvement ≥ 1 From Baseline and no Use of Rescue Therapy at Week 24 | Baseline up to Week 24
Part 1: Proportion of Participants in LGI1 AIE Cohort With mRS Score Improvement ≥ 1 From Baseline and no Use of Rescue Therapy at Week 52 | Baseline up to Week 52
Part 2: Percentage of Participants With Adverse Events (AEs) | From Week 52 up to 2 years

SECONDARY OUTCOMES:
Part 1 (NMDAR AIE Cohort and LGI1 Cohort): Time to mRS Score Improvement ≥ 1 From Baseline Without Use of Rescue Therapy | Baseline up to Week 52
Part 1 (NMDAR AIE Cohort and LGI1 AIE Cohort): Time to Rescue Therapy | Baseline up to Week 52
Part 1 (NMDAR AIE Cohort and LGI1 AIE Cohort): Proportion of Participants With Sustained Seizure Cessation at Week 24 | Baseline up to Week 24
  Sustained seizure cessation is defined as 4 consecutive weeks of no seizures maintained until Week 24 and no use of rescue therapy.
Part 1 (NMDAR AIE Cohort): Change in Clinical Assessment Scale in Autoimmune Encephalitis (CASE) Score From Baseline at Week 24 | Baseline up to Week 24
Part 1 (LGI1 AIE Cohort): Change in CASE Score From Baseline at Week 52 | Baseline up to Week 52
Part 1 (NMDAR AIE Cohort): Montreal Overall Cognitive Assessment (MOCA) Total Score at Week 24 | Baseline up to Week 24
Part 1 (LGI1 AIE Cohort): MOCA Total Score at Week 52 | Baseline up to Week 52
Part 1 (LGI1 AIE Cohort): Rey Auditory Verbal Learning Test (RAVLT) Score at Week 52 | Baseline up to Week 52
Part 1 (NMDAR AIE Cohort): mRS Score at Week 24 (as Measured on a 7-point Scale) | Baseline up to Week 24
Part 1: Percentage of Participants With AEs | Baseline, Week 52, 2 Years
  Severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE V5.0)
Parts 1 and 2: Change from Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline up to 2 years
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (92):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC San Diego, La Jolla, California
  - Hoag Memorial Hospital, Newport Beach, California
  - UCSF- Multiple Sclerosis Centre, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Childrens National Health Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta Center for Advanced Pediatrics, Atlanta, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital Department of Neurology, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - NYU-Langone Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Univ of Pennsylvania Med Ctr, Philadelphia, Pennsylvania
  - University of Texas at Houston, Houston, Texas
  - Swedish Neuroscience Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Ramos Mejía, CABA
  - Hospital Britanico, Ciudad Autonoma Bs As
  - Sanatorio del Sur S.A., San Miguel de Tucumán
- Austria (2):
  - Kepler Universitätsklinikum GmbH - Neuromed Campus, Linz
  - Medizinische Universität Wien, Vienna
- Brazil (5):
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
- China (13):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Beijing Tongren Hospital, Beijing
  - Beijing Tiantan Hospital,Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital - Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Affiliated Hospital of Jining Medical University, Jining
  - Huashan Hospital, Fudan University, Shanghai
  - The First Hospital of Shanxi Medical University, Taiyuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice v Motole, Prague
- Odense Universitetshospital, Neurologisk Afdeling N, Odense C, Denmark
- France (4):
  - Hopital neurologique Pierre Wertheimer - CHU Lyon, Bron
  - Hopital Pitié Salpétrière - CHU, Paris
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - CHRU - Hôpital Bretonneau, Tours
- Komfo Anokye Teaching Hospital, Kumasi, Ghana
- Israel (2):
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - A. O. U. Federico II, Napoli, Campania
  - AOU Seconda Università degli Studi, Napoli, Campania
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
  - AOU Policlinico Giaccone, Palermo, Sicily
- Japan (18):
  - Fujita Health University Hospital, Aichi
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hokkaido University Hospital, Hokkaido
  - Hyogo prefectural Kobe Children's Hospital, Hyogoken
  - Kobe University Hospital, Hyōgo
  - Kagoshima City Hospital, Kagoshima
  - St.Marianna University School of Medicine hospital, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Tohoku University Hospital, Miyagi
  - The University of Osaka Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Ageo Central General Hospital, Saitama
  - Juntendo University Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
- Erasmus MC, Rotterdam, Netherlands
- Poland (4):
  - Regionalny Szpital Specjalistyczny im. W. Bieganskiego, Grudzi?dz
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
  - SPSK nr 1, Zabrze
- National University Hospital (NUH), Singapore, Singapore
- Seoul National University Hospital, Seoul, South Korea
- Spain (3):
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Regional Universitario de Malaga ? Hospital General, Málaga
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, North Dist.
  - Chang Gung Memorial Hospital - Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing